CLINICAL TRIAL: NCT01541163
Title: Assessment of Relationship Between Acute Ischemic Stroke and Heart Disease
Brief Title: Heart and Ischemic STrOke Relationship studY
Acronym: HISTORY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Palacky University (Other)
Responsible Party: Principal Investigator, Michal Kral, Study Director, University Hospital Olomouc
Other Study IDs: NT 11046-6/2010; Grant project No.86-17 (Other: University Hospital Olomouc)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Brain Ischemia; Acute Stroke; Heart Diseases
Keywords: Ischemia; Brain Infarction; Acute Stroke; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Brain Ischemia; Stroke; Heart Diseases; Ischemia; Brain Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Ischemic Stroke: Patients with acute ischemic stroke admitted within 12 hours after onset.

SUMMARY:
Although cardio-embolic etiology of ischemic stroke (IS) is largely respected, there is still no clear recommendation for routine complex cardiological examination in all IS patients. Using complex cardiological examination the investigators expect:

1. more accurate detection of patients with concomitant heart disease (cardiac rhythm disorder, valve disorders, acute coronary syndrome, cardiac thrombus and myxoma, atrial and ventricle septum defects)
2. higher number of etiologically determinated IS, which is crucial for accurate secondary prevention.

DETAILED DESCRIPTION:
The investigators expect significant changes of biochemical parameters (NT pro B-type of natriuretic peptide, pro-atrial natriuretic peptide, creatinkinase MB, troponin T), inflammatory markers (interleukine 6, procalcitonin, high sensitive C-reactive protein), and coagulation parameters in patients with CE IS compared to other causes of IS.

Assessing the glomerular filtration of cystatin C, glycated haemoglobin and serum lipids and its correlation with prior medicament use will allow to evaluate the long-term compensation of arterial hypertension, diabetes mellitus and dyslipidemia in IS patients.

In addition to the above mentioned comprehensive cardiological examinations, 1- and 3-week ECG-Holter will be performed in subpopulation of patients old up to 50 years and with cryptogenic ischemic stroke in the period from 1st May 2013 to 31st December 2015. These patients will also fill in a special epidemiologic questionnaire. Anticipated enrollment in this substudy of HISTORY study is 40 - 80 patients.

In selected young cryptogenic stroke patients, a subcutaneous cardiac monitor was implanted for the detection of paroxysmal atrial fibrillation in the period from 1st January 2014 to 31st December 2015.

From 2016 in young ischemic stroke (IS) patients under 50 years, a standard perfusion/ventilation scintigraphy of lungs will be performed to exclude acute pulmonary embolization (coincidental) in case of elevated serum D-dimers after admission.

In all enrolled young IS patients, a BP Holter will be performed after the discharge home to exclude possible arterial hypertension, which did not presented during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke admitted within 12 hours from stroke onset at stroke center

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive ischemic stroke patients within 12 hours from stroke onset, who will be admitted at Comprehensive Stroke Center, Department of Neurology, University Hospital Olomouc from the October 2010 until December 2015.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
To assess the serum level profile of cardiac troponin T (cTnT) in acute ischemic stroke (AIS) patients and to evaluate factors associated with increased serum level of cTnT. | Within 12 hours after ischemic stroke onset.

SECONDARY OUTCOMES:
Correlation between location and volume of brain infarction. | At admission within 12 hours after stroke onset and after 24hours.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kral, MD, Study Director — University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

REFERENCES:
- [Derived] Franc D, Sanak D, Kral M, Hutyra M, Taborsky M, Divisova P, Zapletalova J. Impact of prior oral anticoagulation on admission stroke severity in patients with atrial fibrillation. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2024 Jul 16. doi: 10.5507/bp.2024.024. Online ahead of print. PMID 39023063
- [Derived] Franc D, Sanak D, Divisova P, Lyskova L, Bartkova A, Zapletalova J, Kral M, Dornak T, Polidar P, Veverka T, Kanovsky P. Socioeconomic status and lifestyle in young ischaemic stroke patients: a possible relationship to stroke recovery and risk of recurrent event. Cent Eur J Public Health. 2021 Sep;29(3):223-229. doi: 10.21101/cejph.a6697. PMID 34623123
- [Derived] Divisova P, Sanak D, Vaclavik J, Kral M, Hutyra M, Zapletalova J, Bartkova A, Franc D, Dornak T, Veverka T, Taborsky M, Kanovsky P. Arterial Hypertension and Risk of Recurrent Event in Young Ischemic Stroke Patients. Can J Neurol Sci. 2021 May;48(3):358-364. doi: 10.1017/cjn.2020.200. Epub 2020 Sep 11. PMID 32912364
- [Derived] Divisova P, Sanak D, Kral M, Bartkova A, Hutyra M, Zapletalova J, Dornak T, Spacek M, Franc D, Polidar P, Veverka T, Kanovsky P. Young cryptogenic ischemic stroke: A descriptive analysis of clinical and laboratory characteristics, outcomes and stroke recurrence. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):105046. doi: 10.1016/j.jstrokecerebrovasdis.2020.105046. Epub 2020 Jun 23. PMID 32807456
- [Derived] Sanak D, Divisova P, Hutyra M, Kral M, Bartkova A, Zapletalova J, Latal J, Dornak T, Hudec S, Franc D, Polidar P, Veverka T, Kanovsky P. Risk of recurrent ischemic stroke in young cryptogenic patients with embolic stroke of undetermined source. J Neurol Sci. 2020 Sep 15;416:116985. doi: 10.1016/j.jns.2020.116985. Epub 2020 Jun 13. PMID 32563078
- [Derived] Sanak D, Hutyra M, Kral M, Bartkova A, Zapletalova J, Fedorco M, Veverka T, Vindis D, Dornak T, Skala T, Skoloudik D, Taborsky M, Kanovsky P. Paroxysmal atrial fibrillation in young cryptogenic ischemic stroke: A 3-week ECG Holter monitoring study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2015 Jun;159(2):283-7. doi: 10.5507/bp.2015.019. Epub 2015 Apr 24. PMID 25916280
- [Derived] Sanak D, Hutyra M, Kral M, Bartkova A, Zapletalova J, Fedorco M, Veverka T, Vindis D, Dornak T, Skala T, Skoloudik D, Taborsky M, Kanovsky P. Atrial fibrillation in young ischemic stroke patients: an underestimated cause? Eur Neurol. 2015;73(3-4):158-63. doi: 10.1159/000369793. Epub 2015 Jan 8. PMID 25573455
- [Derived] Kral M, Sanak D, Veverka T, Hutyra M, Vindis D, Bartkova A, Kuncarova A, Dornak T, Cechakova E, Herzig R, Langova K, Kanovsky P, Skoloudik D. Troponin T: Correlation with location and volume of acute brain infarction. Int J Cardiol. 2015 Feb 15;181:127-32. doi: 10.1016/j.ijcard.2014.12.027. Epub 2014 Dec 3. PMID 25497535
- [Derived] Kral M, Skoloudik D, Sanak D, Veverka T, Bartkova A, Dornak T, Hutyra M, Vindis D, Ulehlova J, Slavik L, Svabova M, Kubickova V, Herzig R, Kanovsky P. Assessment of relationship between acute ischemic stroke and heart disease--protocol of a prospective observational trial. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2012 Sep;156(3):284-9. doi: 10.5507/bp.2012.094. Epub 2012 Oct 4. PMID 23069890
- See also: University Hospital Olomouc — http://www.fnol.cz/
- See also: Ministry of Health of Czech Republic — http://www.mzcr.cz/
- See also: Biomedical Papers - Protocol of a prospective observational trial — http://biomed.papers.upol.cz/pdfs/bio/2012/03/16.pdf
- See also: Kral M et al. Troponin T in Acute Ischemic Stroke. Am J Cardiol. 2013 Jul 1;112(1):117-21. Epub 2013 Apr 6. — http://www.ncbi.nlm.nih.gov/pubmed/23566538